CLINICAL TRIAL: NCT01764217
Title: Predicting Clinical Response and Outcome After Definitive Irradiation With MRI-Guided Adaptive Brachytherapy in Uterine Cervix Cancer
Brief Title: Prediction of Clinical Response and Outcome in Uterine Cervix Cancer
Status: Completed | Type: Observational
Sponsor: Maastricht Radiation Oncology (Other)
Collaborators: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: CERVMA01
Record Dates: First submitted 2012-11-12; First posted 2013-01-09 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Cervix Cancer
Keywords: Cervix Cancer; SUV; Radiotherapy; Outcome Prediction; Imaging; PET
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Observational study based on the routine clinical treatment and diagnostic course, to correlate imaging features with outcome objectives. Outcome will evaluated as clinical response to the standard treatment and as recurrence and survival in the follow up. The study hypothesis is that data extracted form FDG-PETCT used in the routine clinical practice can predict outcomes following standard treatment.

DETAILED DESCRIPTION:
This study will prospectively collect patients undergoing to the standard diagnostic and treatment protocol in Maastro Clinic. Any difference in the normal procedure will be adopted. The aim is to extrapolate form the PET images some features of the metabolic tumor activity to associate with different outcomes and tumor behaviours.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed cervix carcinoma (all subtypes)
* Tumor Stages FIGO IB - IVA
* Scheduled for primary curative radiotherapy (either or not combined with chemotherapy or hyperthermia)
* pre treatment FDG PETCT
* The patient is willing and capable to comply with study procedures
* 18 years or older
* Written informed consent to the treatment

Exclusion Criteria:

* Recent (< 3 months) myocardial infarction
* Uncontrolled infectious disease
* Pregnant or breast feeding and/or not willing to take adequate contraceptive measures during the study
* Previous surgery to the Cervix
* Previous radiation to the Cervix

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Histologically proven cervical uterine cancer, undergoing to conventional radiotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2006-07; Primary Completion 2006-07 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Change of SUV-related tumor characteristics predicting recurrence | Changes of parameters will be calculated on the pretreatment scan, than in average 2.5 months after the last radiotherapy session, than at least each 6 month for the first 2 years, eventually shortening the interval if clinically needed
  * Standard Uptake Value Max (SUV- defined as the ratio of tissue radioactivity concentration (e.g. in MBq/kg=kBq/g) at time t, c(t), and the injected activity ( in MBq) at the time of injection (t=0) divided by the body weight in kg),
  * Metabolic Volume (MV) calculated in cc:volume of the evaluable metabolic activity on the PET scan calculated in a specific Region of Interest (ROI) semiautomatically delineated on the primary tumor in the uterine Cervix

SECONDARY OUTCOMES:
Change of SUV-related tumor characteristics predicting clinical overall response | Changes of parameters will be calculated on the pretreatment scan, and in average 2.5 months after the last radiotherapy session.
  * Standard Uptake Value Max (SUV- defined as the ratio of tissue radioactivity concentration (e.g. in MBq/kg=kBq/g) at time t, c(t), and the injected activity ( in MBq) at the time of injection (t=0) divided by the body weight in kg),
  * Ratio of Pre/Post treatment SUV MAX,
Radiomics Features | Radiomics features will be evaluated on the preteratment CT-fdg PET scan in average at least 2 weeks after the end of the accrual.
  * We will apply a high throughput approach to convert medical images to minable data, where it is hypothesized that it will improve tumor characterization and treatment outcome prediction.
  * Extracted imaging features consist firstly of global properties, providing information on the first order histogram of voxel intensity values within the tumor VOI.
  * Local and regional textural features describing patterns and spatial distribution of voxel intensities, are calculated from respectively gray level co-occurrence and gray level run-length matrix representations. Images will be discretized before texture analysis, which allows for a direct comparison of all calculated textural features between patients. Co-occurrence and gray level run-length matrices are determined considering 26-connected voxels (i.e. voxels were considered to be neighbors in all 13 directions in three dimensions) and a distance of 1 between consecutive voxels. Features derived from the co-occurrence and gray
Interobserver variability of Gross Tumor Volume (GTV) contours | GTV's will be delineated 2 weeks after the end of accrual
  * GTV volume in cc contoured by 5 different observers on pretreatment scan: the difference in cc between each contour obtained will be scored
  * GTV Overlapping fraction rate: the overlapping rate of GTV volume between contours

CONTACTS AND LOCATIONS:
Overall Officials: philippe Lambin, Principal Investigator — Maastro Clinic, The Netherlands
Locations (1):
- Philippe Lambin, Maastricht, Limburg, Netherlands